CLINICAL TRIAL: NCT01021007
Title: Clinical Research Study Efficacy of a Prototype Oral Rinse
Acronym: Quigley
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-1007-GIN-02-RR
Record Dates: First submitted 2008-09-26; First posted 2009-11-26 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-10

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Iodine; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): control mouthrinse
  Interventions: Other: water
- B (Experimental): new prototype mouthrinse
  Interventions: Drug: Iodine

INTERVENTIONS:
Drug: Iodine — Rinse 2 times per day for 6 weeks
  Other Names: Iocide (proprietary company name)
  Arms: B
Other: water — Use 2 times per day for 6 weeks
  Other Names: No actives present in control mouthrinse. (Flavored water)
  Arms: A

SUMMARY:
Evaluate the efficacy of an oral rinse on dental plaque and gingival inflammation

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers 18-65 years of age
2. Good general health
3. Must sign informed consent form
4. Minimum of 16 natural uncrowned teeth (excluding third molars) must be present.
5. No history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study.
6. Dental Selection Criteria: Gingivitis patients with a minimum of 16 gradable teeth with a minimum of 6 sites with a GI score of ≥ 3. Subjects will be stratified according to gingivitis severity. Average full mouth GI score should be in the range of 2.0 - 2.5. heavy plaque formers should be avoided. Target a full mouth PI (Quigley-Hein) to be in the range of 1.5-3.0

Exclusion Criteria:

1. Subjects unable or unwilling to sign the informed consent form.
2. Medical condition which requires pre-medication prior to dental visits/procedures
3. Moderate or advanced periodontal disease
4. History of allergy to iodine
5. History of thyroid disease
6. History of diabetes
7. 2 or more decayed untreated dental sites at screening.
8. Other disease of the hard or soft oral tissues.
9. Impaired salivary function (e.g. Sjogren's syndrome or head and neck irradiation).
10. Use of medications that are currently affect salivary flow.
11. Use of antibiotics or antimicrobial drugs within 30 days prior to study visit #1.
12. Pregnant or nursing women.
13. Participation in any other clinical study within 1 week prior to enrollment into this study.
14. Use of tobacco products
15. Subjects who must receive dental treatment during the study dates.
16. Current use of Antibiotics for any purpose.
17. Presence of an orthodontic appliance.
18. History of allergy to common dentifrice ingredients
19. Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)
20. Women of childbearing potential and not on birth control (Diaphragm, birth control pills or implants, IUD (Intrauterine device), condoms).
21. Smoker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cronin, DMD, Principal Investigator
Locations (1):
- New Institutional Service Company, Northfield, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At clinical site
Groups:
- Negative Control Rinse: Placebo mouthrinse
- Iocide Mouthrinse: Experimental mouthrinse
Period: Overall Study
Arm/Group | Negative Control Rinse | Iocide Mouthrinse
Started | 36 | 37
Completed | 34 | 33
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Control Rinse | Iocide Mouthrinse | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 37 | 73
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.8 (8.3) | 36.6 (10.9) | 37.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 53
  Male | 7 | 13 | 20
Region of Enrollment [Number; unit: participants]
  United States | 36 | 37 | 73

OUTCOME MEASURES:

1. Primary Outcome: Gingival Index
Description: 1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Negative Control Rinse | Iocide Mouthrinse
Number analyzed (Participants) | 34 | 33
Units on a scale | 1.90 (0.19) | 1.84 (0.23)
Statistical Analysis 1: Comparison: Negative Control Rinse vs Iocide Mouthrinse; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.005, ANCOVA; ANCOVA method using treatment as the factor and the baseline score as a covariate

2. Primary Outcome: EIBI Bleeding Score: Eastman Indterdental Bleeding Index Scale
Description: 0 = no bleeding or 1=spontaneous bleeding. Both upper and lower gums around each tooth in the mouth are checked for bleeding sites . The total number of 0 & 1 scores are added together and then divided by the total number of sites in the mouth evaluated to give the average number of bleeding sites in the mouth.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: bleeding sites
Arm/Group | Negative Control Rinse | Iocide Mouthrinse
Number analyzed (Participants) | 34 | 33
bleeding sites | 40.82 (16.93) | 34.91 (23.83)
Statistical Analysis 1: Comparison: Negative Control Rinse vs Iocide Mouthrinse; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA; ANCOVA method using treatment as the factor and the baseline score as a covariate

3. Primary Outcome: Plaque Index (Quigley-Hein Score)
Description: Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Negative Control Rinse | Iocide Mouthrinse
Number analyzed (Participants) | 34 | 33
Units on a scale | 2.47 (0.61) | 2.11 (0.70)
Statistical Analysis 1: Comparison: Negative Control Rinse vs Iocide Mouthrinse; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA; ANCOVA method using treatment as the factor and the baseline score as a covariate

ADVERSE EVENTS:
Time Frame: 7 week study period
Arm/Group | Negative Control Rinse | Iocide Mouthrinse
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 12/34 | 9/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Negative Control Rinse (N=34) | Iocide Mouthrinse (N=33)
discomfort in mouth or body (Social circumstances) | 8 (8) | 0 (0) — 1 panelist reported discomfort from a popcorn kernel stuck between teeth. 7 panelists reported discomfort in ranging from a tooth ache to muscle pains. All unrelated to study product use and went away with no lingering effects to the panelist.
Tooth staining (General disorders) | 1 (1) | 7 (7) — Panelist reports the appearence of yellow to brown staining of their teeth. All staining was removed after a dental cleaning. No lingering effects to the panelist.
slight swelling or inflammation of the gums (General disorders) | 3 (3) | 2 (2) — panelists reported slight iritation or tenderness or swelling or inflammation of the tongue or gums. All chages reported to the panelists oral health were resolved during the study and no lingering effects were noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days